CLINICAL TRIAL: NCT00555802
Title: The Effect of Motor Control Exercise Versus General Exercise on Lumbar Local Stabilizing Muscles Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 86-1534
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2007-11

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Motor Control Exercise; General exercise; Ultrasonography, Multifidus; Transversus abdominis; Randomized Controlled trial.
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: exercise — exercise
  Other Names: training

SUMMARY:
The purpose of this study was to evaluate the efficacy of motor control exercises. For this, before and after motor control and general exercises, we determined transverses abdominis and multifidus thickness, activity limitation and pain. We hypothesized that the motor control exercises would increase transverses abdominis and multifidus muscles thickness. Activity limitation and pain would decrease following two protocols that it was more in motor control group than general one.

DETAILED DESCRIPTION:
Musculoskeletal disorders, of which back pain accounts for more than half the number of cases, are the most common cause of chronic incapacity in industrialized countries. Approximately 10-20 percent of patients with low back pain develop chronic pain, defined as low back pain persisting more than 3 months. Low back pain represents a particularly costly sociomedical problem because of the expenditure associated with repeated treatment and the long-term absence from work and need for social support. These patients use more than 80% of health care resources for back problems, and treatment has a low success rate. Thus, the development of effective interventions aimed at management of the chronic problems is urgently required.

Review of studies showed that the effectiveness of stabilization exercises in patients with nonspecific LBP is not yet fully established. In clinical trials that improvement reported after motor control exercise, other intervention accompanied with these exercises. Also, the results of motor control exercise studies are different. On the other hand, the evidence underpins the primary aim of motor control exercise, which is to re-establish normal control of the deep spinal muscles, reducing the activity of more superficial muscles that tend to stiffen the spine and have increased activity in low back pain, and then maintain normal control during progressively more demanding physical and functional tasks. For these reasons, we decided to identify the efficacy of motor control exercises, usually considered as specific trunk muscle stabilization exercises. A randomized controlled trial was only way for identifying the role of these exercises in treating chronic low back pain. Also, our choice coincides with the research agenda set by the 2004 European Guideline.

ELIGIBILITY:
Inclusion Criteria:

* nonspecific low back pain with or without leg pain of at least 3 months duration
* currently seeking care for low back pain
* aged greater than 18 and less than 80 years
* suitable for motor control exercise based on clinical assessment
* The patients must also have sufficient knowledge of the Persian language to understand instructions

Exclusion Criteria:

* suspected or confirmed serious spinal pathology (fracture, metastatic, inflammatory or infective diseases of the spine, cauda equine syndrome, widespread neurological disorder)
* suspected or confirmed pregnancy
* nerve root compromise (2 of strength, reflex or sensation affected for same nerve root)
* spinal surgery
* any of the contraindications to exercise listed on page 42 of the ACSM guidelines

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-04; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Before and after intervention, we assessed the multifidus and abdominal muscles thickness (mm) using a 7.5 MHz B-mode transducer ultrasound, pain through visual analog scale and activity limitation through Back Performance Scale. | Baseline, 16 weeks

SECONDARY OUTCOMES:
Weight, Age, height,BMI,Current duration of pain,Time since first onset | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Akbari, Principal Investigator — Deputy of research, Zahedan university of medical scinces
Locations (1):
- Dept. of physiotherapy, Zahedan university of medical scinces, Zahedan, Sistan & Bladchestan, Iran

REFERENCES:
- [Background] Maher CG, Latimer J, Hodges PW, Refshauge KM, Moseley GL, Herbert RD, Costa LO, McAuley J. The effect of motor control exercise versus placebo in patients with chronic low back pain [ACTRN012605000262606]. BMC Musculoskelet Disord. 2005 Nov 4;6:54. doi: 10.1186/1471-2474-6-54. PMID 16271149
- See also: Spine-health.com has organized its peer-reviewed articles and patient information into Health Hubs dedicated to specific conditions, treatments, and pain management topics. — http://www.spine-health.com